CLINICAL TRIAL: NCT01469091
Title: Tobacco's Impact on Postoperative Complications in Acute Vascular Surgery. A Randomized Clinical Trial
Brief Title: Tobacco's Impact on Postoperative Complications in Acute Surgery
Acronym: ROC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of patient inclusion
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Mette Kehlet, Principal Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Roc-2010
Record Dates: First submitted 2011-10-27; First posted 2011-11-10 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Vascular Disease
Keywords: Acute admittance; Current smoker
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smoking intervention, Nicotine replacement therapy. (Active Comparator)
  Interventions: Behavioral: Smoking intervention.
- Controlgroup (No Intervention)

INTERVENTIONS:
Behavioral: Smoking intervention. — Nicotine replacement therapy and meetings with nurse specialized in smoking intervention.
  Arms: Smoking intervention, Nicotine replacement therapy.

SUMMARY:
The purpose of the study is to see whether intensive smoking intervention on the day of operation can reduce per- and postoperative complications in patients operated for acute ischaemic disease compared to control group with no intervention.

ELIGIBILITY:
Inclusion Criteria:

* acute admittance in a vascular department
* current smoker
* surgery within 7 days
* informed/written consent

Exclusion Criteria:

* alcohol intake > 35 units pr. week
* dementia or mental disease
* > 90 years

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-09 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Postoperative complications. | After 3 months.

SECONDARY OUTCOMES:
SF-36 | After 3 months.
  Patients self-assessed health status.

CONTACTS AND LOCATIONS:
Locations (1):
- Vascular Clinic RK, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Kehlet M, Heeseman S, Tonnesen H, Schroeder TV. Perioperative smoking cessation in vascular surgery: challenges with a randomized controlled trial. Trials. 2015 Oct 5;16:441. doi: 10.1186/s13063-015-0965-x. PMID 26438129